CLINICAL TRIAL: NCT03683914
Title: Vaginal Dinoprostone Prior to Diagnostic Office Hysteroscopy in Postmenopausal Patients: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Vaginal Dinoprostone Prior to Diagnostic Office Hysteroscopy in Postmenopausal Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vaginal dinoprostone
Record Dates: First submitted 2018-09-22; First posted 2018-09-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Office Hysteroscopy
MeSH Terms: interventions — Dinoprostone; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone arm (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: Dinoprostone 3Mg Vaginal Tablet
- placebo (Placebo Comparator): one tablet of placebo inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: placebo vaginal tablet

INTERVENTIONS:
Drug: Dinoprostone 3Mg Vaginal Tablet — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the patient 12 hours before the scheduled office diagnostic hysteroscopy.
  Arms: dinoprostone arm
Drug: placebo vaginal tablet — 1 vaginal tablet of placebo inserted by the patient 12 hours before the scheduled office diagnostic hysteroscopy.
  Arms: placebo

SUMMARY:
To compare the effectiveness of vaginal dinoprostone with placebo in minimising the pain experienced by postmenopausal patients during diagnostic ofﬁce hysteroscopy and to assess the ease of insertion of hysteroscope as reported by the hysteroscopist.

DETAILED DESCRIPTION:
hysteroscopy is commonly used in the diagnosis and treatment of intrauterine lesions such as polyps, ﬁbroids, septa, and adhesions, and in the presence of abnormal bleeding and during the removal of an intrauterine device or foreign body.Cervical ripening is made possible by the use of medication through different routes.The most commonly used agent is misoprostol,a synthetic prostaglandin E1 (PGE1) analogue that is frequently administered in off-label use in obstetrics and gynaecology for medical abortion, labor induction, endometrial biopsy, dilatation and curettage, intrauterine device insertion, myomectomy, postpartum haemorrhage, and cervical ripening.In contrast, dinoprostone, a natural PGE2, is mostly used in obstetrics for cervical ripening and the stimulation of uterine contractions to induce labor.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients with an indication for ofﬁce hysteroscopy (postmenopausal bleeding or abnormal ultrasound ﬁndings)

Exclusion Criteria:

* • Nulliparous patients

  * patients with cervical pathology
  * retroverted uterus (detected by transvaginal ultrasound)
  * previous cervical surgery
  * patients with severe vaginal bleeding
  * allergy or contraindications to dinoprostone therapy (asthma, liver, kidney, or heart disease).

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | an expected average of 10 minutes
  Pain intensity will be assessed by visual analogue scale during the procedure.visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Intensity of pain | 30 minutes after the procedure
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure.visual analogue scale ranging from 0 to 10
Operative time | an expected average 10 minutes
  From the introduction of hysteroscope into the vagina till compilation of hysteroscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt